CLINICAL TRIAL: NCT05419141
Title: A Prospective Study on Accuracy and Safety of Coplanar Template Assisted CT-guided Pelvic and Groin Areas Biopsy
Brief Title: Accuracy of Coplanar Template Assistance for Pelvic and Groin Areas Biopsy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Qiu Bin, Principal Investigator, Peking University Third Hospital
Other Study IDs: ChiECRCT20220127
Record Dates: First submitted 2022-06-10; First posted 2022-06-15 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Pelvic and Groin Areas Biopsy
Keywords: Pelvic; Groin; Biopsy; Coplanar template.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In recent years, template guidance has been applied and developed in the field of puncture related operations, such as template-assisted radioactive seed implantation. With the guidance of template, needle pathway of seed implantation, biopsy and fiducial marker implantation can be precisely planned

, which is conducive to accurate proceeding. Templates can be divided into coplanar templates and non-coplanar templates. The digital coplanar template coordinate puncture system has been developed in China and has been applied in clinical practice. In our previous studies, coplanar template assisted CT-guided radioactive seed implantation has good clinical feasibility for percutaneous biopsy of small pulmonary nodules. However, the accuracy of coplanar template assistance for abdominal tumor puncture are lacking in prospective studies. The study aims to prospectively observe the accuracy and safety of coplanar template assisted CT-guided Pelvic and Groin Areas biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 18 to 90
2. Single or multiple Pelvic and Groin Areas mass (solid, partially solid)
3. Without taking drugs affecting coagulation and/or platelet aggregation are used; If used, the drug has been discontinued for a sufficient period of time (e.g. 1 week)

   - Page 3 of 4 [DRAFT] -
4. KPS>60 points, no serious or uncontrolled underlying diseases, clinical evaluation patients can tolerate puncture
5. Planned biopsy with applicable puncture path
6. With informed consent.

Exclusion Criteria:

-

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 1. Poor organ function (e.g. lung function FEV1<40% and/or DLCO<50%)
  2. The lesion close to blood vessels and intestine, or there is portal vein hypertension and superior vena cava compression, etc., which are expected to have high risks of puncture bleeding and intestinal injury
  3. Poor compliance and unable to complete coordination
  4. Paticipant who is considered inappropriate or unwilling to participate in this clinical trial for other reasons.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2024-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Depth | during the operation
  Depth (millimeter) difference between actual puncture and planned puncture pathway
Accuracy of Angle | during the operation
  Angle (degree) difference between actual puncture and planned puncture pathway

SECONDARY OUTCOMES:
Success rate of needle puncture | during the operation
  Success rate of needle puncture
Complication rate | perioperative the operation
  such as pneumoperitoneum, subcutaneous emphysema, hemorrhage, infection, etc.
operating duration | during the operation
  operating duration from the starting to the ending
Number of CT scans | during the operation
  Number of CT scans

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - Bin Qiu, M.D., Beijing

IPD SHARING:
Plan to Share IPD: Undecided